CLINICAL TRIAL: NCT05380960
Title: A Study on the State of Coagulability in Patients With Chronic Obstructive Disease Admitted to Assiut University Hospital
Brief Title: Blood Hpercoagublity in Copd
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Zeinab Nashaat Mohamed Omar, hpercoagubility in copd, Assiut University
Other Study IDs: hpercoagubiliy in copd
Record Dates: First submitted 2022-05-14; First posted 2022-05-19 (Actual); Last update posted 2022-05-19 (Actual); Status verified 2022-05

CONDITIONS: Blood Coagulability in Copd

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- copd in acute excerbtion: (1) The first group (COPD group) in acute exacerbaction: We plan to include COPD patients who will be admitted to the Chest Diseases Department with severe exacerbation requiring admission to the RICU (severe dyspnea that responds inadequately to initial emergency therapy, changes in mental status, persistent or worsening hypoxemia, persistent or worsening respiratory acidosis, the need for ventilatory support, and/or hemodynamic instability.
  Interventions: Device: cbc coaglation profile
- (2) The second group (non-COPD lung diseases group).: We plan to include patients admitted at the RICU with bronchial asthma, bronchiectasis, pneumonia, and interstitial lung disease.
  Interventions: Device: cbc coaglation profile
- normal persons: have no diseases
  Interventions: Device: cbc coaglation profile

INTERVENTIONS:
Device: cbc coaglation profile — The Demographic, clinical, and laboratory data for the enrolled subjects will be collected. To assess the coagulability state in the participants, we will measure the levels of certain markers in the blood that are thought to be associated with an increased coagulability. A comparison will be made between the different included groups regarding the level of these markers. These markers included complete blood count (CBC) indices (hematocrit, red cell distribution width, platelets count, mean platelet volume and platelet distribution width), C - reactive protein, d dimer, and blood coagulation tests (prothrombin time, international normalized ratio and partial thromboplastin time).
  Other Names: d dimer crp

SUMMARY:
"The objective of this study is to evaluate the blood coagulability state in patients with COPD admitted at Assiut University Hospital"

DETAILED DESCRIPTION:
Chronic Obstructive Pulmonary Disease (COPD) is a chronic debilitating lung disease with a high prevalence of approximately 380 million cases worldwide [1]. It is currently the third leading cause of death, responsible for approximately 6% of the world's total deaths (approximately 3.3 million annually) [2]. In addition to the known devastating respiratory consequences, a large number of studies support the hypothesis that COPD increases the risk for both venous thromboembolism (VTE) and cardiovascular disease (CVD) Although the observed association of COPD with CVD and VTE can be partially explained by comorbidities and shared risk factors, there is strong evidence that COPD increases the risk for cardiovascular morbidity and mortality independently of age, gender, and smoking history [3,4]. It is of note that up to 63.5% of patients with COPD die of comorbid circulatory system diseases [5].

Increased thrombin formation [6] , reflected by elevated thrombin-antithrombin com- plexes [7] , tissue factor procoagulant activity [8] and activated factor XI [9] , increased d-dimers [10] , and FI [11] , FII and FX [12] levels in the serum of COPD patients support the theory that a hypercoagulable state occurs in patients with COPD and might contribute to the incidence of atherothrombotic events and VTE, increasing disease related morbidity and mortality.

Potential pathways illustrating pathogenetic mechanisms of increased risk of CVD and VTE in COPD are imprecise. Evidence illustrates four possible synergistic mechanisms: systemic inflammation [13], platelet activation [14] , oxidative stress [15], and hypoxia, either sustained in severe COPD or intermittent during exercise and sleep [16,17]

ELIGIBILITY:
Inclusion Criteria:

1. The first group (COPD group) in acute exacerbaction: We plan to include COPD patients who will be admitted to the Chest Diseases Department with severe exacerbation requiring admission to the RICU (severe dyspnea that responds inadequately to initial emergency therapy, changes in mental status, persistent or worsening hypoxemia, persistent or worsening respiratory acidosis, the need for ventilatory support, and/or hemodynamic instability.

   The diagnosis of COPD was based on the patient's medical history obtained from the patient himself and/or the family of the patient, consistent physical findings, previous spirometry and/or evidence of hyperinflation on current or previous chest radiograph.

   The participants will be divided into three groups:
2. The second group (non-COPD lung diseases group). We plan to include patients admitted at the RICU with bronchial asthma, bronchiectasis, pneumonia, and interstitial lung disease.
3. The the third group (healthy control group). This group will include volunteers who are apparently healthy in every aspect exculsion ctritria 1. Primary hematological disease. 2. Coagulation disorders. 3. Malignancy anywhere in the body. 4. Hepatic disease. 5. Renal disease. 6. Taking anticoagulant and/or antiplatelet medications

Exclusion Criteria:

-

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: 1. The first group (COPD group) in acute exacerbaction: We plan to include COPD patients who will be admitted to the Chest Diseases Department with severe exacerbation requiring admission to the RICU (severe dyspnea that responds inadequately to initial emergency therapy, changes in mental status, persistent or worsening hypoxemia, persistent or worsening respiratory acidosis, the need for ventilatory support, and/or hemodynamic instability.
     The diagnosis of COPD was based on the patient's medical history obtained from the patient himself and/or the family of the patient, consistent physical findings, previous spirometry and/or evidence of hyperinflation on current or previous chest radiograph.
     The participants will be divided into three groups:
  2. The second group (non-COPD lung diseases group). We plan to include patients admitted at the RICU with bronchial asthma, bronchiectasis, pneumonia, and interstitial lung disease.
  3. The the third group (healthy control group)
Sampling Method: Non-Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2022-06-01 (Estimated); Primary Completion 2023-09-01 (Estimated); Study Completion 2023-12-01 (Estimated)

PRIMARY OUTCOMES:
"The objective of this study is to evaluate the blood coagulability state in patients with COPD admitted at Assiut University Hospital" | baseline
  The Demographic, clinical, and laboratory data for the enrolled subjects will be collected. To assess the coagulability state in the participants, we will measure the levels of certain markers in the blood that are thought to be associated with an increased coagulability. A comparison will be made between the different included groups regarding the level of these markers. These markers included complete blood count (CBC) indices (hematocrit, red cell distribution width, platelets count, mean platelet volume and platelet distribution width), C - reactive protein, d dimer, and blood coagulation tests (prothrombin time, international normalized ratio and partial thromboplastin time).

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Castellana G, Intiglietta P, Dragonieri S, Carratu P, Buonamico P, Peragine M, Capozzolo A, Carone M, Carpagnano GE, Resta O. Incidence of deep venous thrombosis in patients with both Pulmonary Embolism and COPD. Acta Biomed. 2021 Jul 1;92(3):e2021210. doi: 10.23750/abm.v92i3.11258. PMID 34212912
- [Background] Jimenez D, Agusti A, Tabernero E, Jara-Palomares L, Hernando A, Ruiz-Artacho P, Perez-Penate G, Rivas-Guerrero A, Rodriguez-Nieto MJ, Ballaz A, Aguero R, Jimenez S, Calle-Rubio M, Lopez-Reyes R, Marcos-Rodriguez P, Barrios D, Rodriguez C, Muriel A, Bertoletti L, Couturaud F, Huisman M, Lobo JL, Yusen RD, Bikdeli B, Monreal M, Otero R; SLICE Trial Group. Effect of a Pulmonary Embolism Diagnostic Strategy on Clinical Outcomes in Patients Hospitalized for COPD Exacerbation: A Randomized Clinical Trial. JAMA. 2021 Oct 5;326(13):1277-1285. doi: 10.1001/jama.2021.14846. PMID 34609451
- [Background] Couturaud F, Bertoletti L, Pastre J, Roy PM, Le Mao R, Gagnadoux F, Paleiron N, Schmidt J, Sanchez O, De Magalhaes E, Kamara M, Hoffmann C, Bressollette L, Nonent M, Tromeur C, Salaun PY, Barillot S, Gatineau F, Mismetti P, Girard P, Lacut K, Lemarie CA, Meyer G, Leroyer C; PEP Investigators. Prevalence of Pulmonary Embolism Among Patients With COPD Hospitalized With Acutely Worsening Respiratory Symptoms. JAMA. 2021 Jan 5;325(1):59-68. doi: 10.1001/jama.2020.23567. PMID 33399840
- [Background] Lankeit M, Held M. Incidence of venous thromboembolism in COPD: linking inflammation and thrombosis? Eur Respir J. 2016 Feb;47(2):369-73. doi: 10.1183/13993003.01679-2015. No abstract available. PMID 26828045